CLINICAL TRIAL: NCT06830694
Title: Clinical Trial for Safety and Effectiveness Evaluation of Tarlatamab (AMG757) with Etoposide, Carboplatin and Atezolizumab in Transformed Small Cell Lung Cancer Patients from Adenocarcinoma After EGFR TKI Treatment: Phase II Multicenter Clinical Trial
Brief Title: Clinical Trial for Safety and Effectiveness Evaluation of Tarlatamab (AMG757) with Etoposide, Carboplatin and Atezolizumab in Transformed Small Cell Lung Cancer Patients from Adenocarcinoma After EGFR TKI Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Myung-Ju Ahn (Other)
Responsible Party: Sponsor-Investigator, Myung-Ju Ahn, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01-014
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Carcinoma of Lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): * Concomitant Chemotherapy Phase: for 4 cycles Q3W Cycle 1 (21-day cycle): Atezolizumab 1200 mg IV followed by carboplatin to match AUC 5.0 IV on day 1 and then etoposide 100 mg/m2 IV on day 1- day 3.
  * Maintenance Tarlatamab Q2W plus Atezolizumab Q4W Cycle 5 (28-day cycle): Atezolizumab 1200 mg IV Q4W on day 1 followed by tarlatamab 1mg IV on day 1 and 10mg IV on day 8 and Day 15 in the maintaining setting. From C6 Atezolizumab 1200 mg IV Q4W on day 1 followed by tarlatamab 10mg IV on day 1 and day 15 will be applied.
  Interventions: Drug: Atezolizumab, Etoposide, Carboplatin, Tarlatamab

INTERVENTIONS:
Drug: Atezolizumab, Etoposide, Carboplatin, Tarlatamab — Cycle 1~4 : Atezolizumab 1200 mg IV, carboplatin AUC 5.0 IV, Etoposide 100 mg/m2 IV Cycle 5~ : Atezolizumab 1200 mg IV, Tarlatamab 1 or 10mg IV

SUMMARY:
The primary treatment option for non-small cell lung cancer (NSCLC) adenocarcinoma (ADC) with activating epidermal growth factor receptor (EGFR) mutation is EGFR tyrosine kinase inhibitor (TKI). After a certain period of treatment with EGFR TKI, acquired resistance emerges most frequently with a secondary mutation, p.T790M (36-50%), followed by MET amplification (10-19%). Interestingly, up to 3-5% of patients experience histological transformation into small cell lung cancer (SCLC).

As an underlying mechanism, ADC with a predisposed clonally inactivated Rb and p53 mutation and APOBEC mutation signature is known to be associated with SCLC transformation. The transformed SCLC harbors similar morphological and immunohistochemical (IHC) characteristics as those observed in de novo SCLC, including high expression of chromogranin and synaptophysin. However, little is known about the clinical outcomes of transformed SCLC, with limited studies arguing that their outcomes are similar to those of de novo SCLC, where the median overall survival is approximately 9 to 10 months after the transformation.

As the first line treatment of SCLC, atezolizumab or durvalumab with four cycles of conventional chemotherapy followed by maintenance therapy demonstrated prolonged overall survival (OS) and placed as the standard treatment option. However, median progression-free survival (PFS) of both study was only 5.2 months and 5.1 months, despite the objective response rate showing 60.2% and 79%. This finding suggest further development of maintenance treatment strategy to prolonged longer duration of response to the treatment.

In addition to the conventional treatment, Tarlatamab (AMG757), bispecific t-cell engager (BiTE), designed to engage DLL3 on SCLC and CD3 on T-cell has been tested in SCLC. DLL3 is expressed in more than 80% of patients with SCLC, regardless of disease stage and researched for the potential target protein for the antibody based treatment in SCLC. By targeting DLL3 using Tarlatamab, engagement of tumor antigen and CD3 lead to cytotoxic synapse formation, triggering the release of proinflammatory cytokines, perforin, and granzymes from activated T-cells, potentially resulting apoptosis. The first clinical outcome of Tarlatamab was reported from the DeLLphi-300 study, phase 1 dose exploration study, showing confirmed partial response in 23% of the heavily treated SCLC and 37% of the patients showed decrease in tumor burden. Median duration of response was 13.0 months (95% confidential interval CI: 6.2 - 14.9 months), median PFS of 3.7 months and median OS was 13.2 months. In the treatment naïve SCLC, DeLLphi-303 study, phase 1b study combining tarlatamab + PD-L1 inhibitor + carboplatin and etoposide, is ongoing to evaluate the clinical efficacy in the front line setting which include only histologically confirmed extensive disease SCLC population (NCT05361395).

Based on previous clinical and pre-clinical outcomes, showing similar disease characteristics between transformed SCLC from the adenocarcinoma who treated with EGFR TKI with de novo SCLC, this study is designed to evaluate the clinical efficacy of tarlatamab with currently standard treatment in transformed SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed SCLC and no prior systemic treatment for SCLC
2. Patient initially diagnosed with activating EGFR mutation (L858R, Del 19) and treated with any kind of EGFR TKI.
3. Confirmed SCLC transformation right after EGFR TKI treatment failure.
4. Age ≥19 years
5. ECOG performance status of 0 to 1
6. Had at least one measurable lesion.
7. Adequate organ function

   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL
   * Estimated glomerular filtration rate based on Modification of Diet in Renal Disease calculation > 30 mL/min/1.73 m2
   * Aspartate aminotransferase and alanine aminotransferase ≤ 3 x upper limit of normal (ULN) (or ≤ 5 x ULN for subjects with liver involvement)
   * Total bilirubin ≤ 1.5 x ULN (or ≤ 2 x ULN for subjects with liver metastases)
   * Prothrombin time (PT)/international normalized ratio and partial thromboplastin time or activated partial thromboplastin time ≤ 1.5 x institutional ULN Note: Subjects on stable anticoagulation therapy are allowed.
8. Pulmonary function: No clinically significant pleural effusion at the timepoint of screening. Pleural effusion with no significant symptom is allowed for enrollment.
9. Cardiac function: Cardiac ejection fraction ≥ 50%
10. Female subjects must either be of non-reproductive potential
11. Female subject with reproductive potential can be enrolled with agreement to following guidance.

    * subject uses contraception during treatment and through 60 days after receiving last dose of tarlatamab or for 6 months after last dose of carboplatin and/or etoposide and 5 months after last dose of atezolizumab.
12. Subject is willing and able to comply with the protocol
13. Signed written informed consent

Exclusion Criteria:

1. Treated with additional chemotherapy after confirmed with transformed SCLC.
2. Previously exposed to the immune checkpoint inhibitor treatment.
3. Untreated symptomatic brain metastases or leptomeningeal disease.

   * Asymptomatic brain metastases can be enrolled per investigator decision
4. Uncontrolled systemic illness including uncontrolled hypertension, active bleeding, or active infection.
5. Past medical history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonitis which required steroid treatment, active non- infectious pneumonitis
6. Active or prior documented autoimmune or inflammatory disorders
7. Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 6 months prior to first dose of study treatment
8. History of solid organ transplant.
9. Major surgical procedures within 28 days prior to first dose of study treatment.
10. History of allergic reactions or acute hypersensitivity reactions to antibody therapies, platinum chemotherapy, or etoposide.
11. Disagree to the guidance of contraception during the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | Up to 6months

SECONDARY OUTCOMES:
Objective response rate(ORR) | About 36 months
Duration of response(DOR) | About 36 months
Overall survival(OS) | About 36 months